CLINICAL TRIAL: NCT02451020
Title: Acclimatization of Healthy Subjects During a Stay at 3200 m
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK15-2015_V2
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Effects of High Altitude
Keywords: healthy volunteers; acclimatization; sleep; hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altitude exposure (Experimental): Stay at 3200 m for 3 weeks
  Interventions: Other: Altitude exposure

INTERVENTIONS:
Other: Altitude exposure — Participants will stay for 3 weeks at an altitude of 3200 m

SUMMARY:
The study evaluates respiratory acclimatization in healthy lowlanders staying for 3 weeks at 3200 m.

DETAILED DESCRIPTION:
This study evaluates the effect of 3 weeks altitude acclimatization on sleep related breathing disturbances in healthy subjects staying at 3200 m. Participants living in Bishkek, Kyrgyzstan (700 m), will be transferred by car within 4 h to the Tuja Ashu high altitude clinic (3200 m). Outcomes will be assessed repeatedly during the stay at 3200 m.

ELIGIBILITY:
Inclusion Criteria:

* Perfect health
* Born, raised and currently living at low altitude (<800m)
* Informed consent.

Exclusion Criteria:

* Any acute or chronic disease
* heavy smoking (>20 cigarettes per day).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2015-08-09 (Actual); Study Completion 2015-08-09 (Actual)

PRIMARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | night 7 at 3200 m
  Difference in mean nocturnal oxygen saturation between night 1 and night 7

SECONDARY OUTCOMES:
Mean nocturnal oxygen saturation measured by pulse oximetry | night 1 at 3200 m
  Difference in mean nocturnal oxygen saturation between night 1 at 3200 and night 1 at 700 m
Mean nocturnal oxygen saturation measured by pulse oximetry | night 21 at 3200 m
  Difference in mean nocturnal oxygen saturation between night 21 and night 1 at 3200 m
Mean nocturnal oxygen saturation measured by pulse oximetry | night 1 at 700 m (low altitude baseline)
  Mean nocturnal oxygen saturation during night 1 at 700 m

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich; Talant M Sooronbaev, MD, Study Director — National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan
Locations (1):
- National Center of Cardiology and Internal Medicine, Bishkek, Kyrgyzstan